CLINICAL TRIAL: NCT07395856
Title: A Study on the Involvement of Rosa Roxburghii in Oxidative Stress in Knee Osteoarthritis and Its Impact on Rehabilitation of Patients After Total Knee Arthroplasty
Brief Title: A Study on Rosa Roxburghii for Knee Replacement Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shuguang Gao (Other)
Responsible Party: Sponsor-Investigator, Shuguang Gao, Prof., Xiangya Hospital of Central South University
Organization: Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYH20250018
Record Dates: First submitted 2026-01-09; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis
Keywords: Rosa roxburghii; Total Knee Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosa roxburghii (Experimental)
  Interventions: Dietary Supplement: Rosa roxburghii
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Rosa roxburghii — Enrolled patients will take 3g of Rosa roxburghii juice freeze-dried powder dissolved in 400-500ml of warm water with breakfast daily, starting from the day after surgery and continuing for 30 consecutive days.
  Arms: Rosa roxburghii
Other: Placebo — Starting from the first postoperative day, patients take placebo 3g/day after breakfast, dissolved in 200ml of warm water (40-50°C), for 4 consecutive weeks.
  Arms: placebo

SUMMARY:
This clinical trail is to investigates the effect of Rosa roxburghii juice freeze-dried powder on the recovery of patients undergoing total knee arthroplasty due to knee osteoarthritis. The participants are divided into an experimental group and a placebo group. Enrolled patients will take 3g of Rosa roxburghii juice freeze-dried powder or a placebo dissolved in 400-500ml of warm water with breakfast daily, starting from the day after surgery and continuing for 30 consecutive days. Data on inflammatory markers, oxidative stress indicators, and knee function scores will be collected from the participants one day before surgery, as well as on the first, third, and thirtieth days after surgery.

DETAILED DESCRIPTION:
Cohort Setting: Two cohorts: Intervention group (TTRJ group) receiving standard postoperative rehabilitation plus freeze-dried RRTJ juice powder; Control group receiving standard postoperative rehabilitation plus an equal dose of placebo.

Perioperative Management:

1. Anesthesia: All patients receive postoperative analgesia education and VAS scale training one day preoperatively and sign informed consent. Routine fasting for 12 hours preoperatively. Upon entering the operating room, venous access is established, and ECG, non-invasive blood pressure, and pulse oximetry are monitored. General anesthesia is used.
2. Surgical Procedure: TKA via anterior midline approach. After incising the deep fascia, the patella is everted to expose the joint surfaces. Hyperplastic synovium within the joint cavity is excised, preserving the infrapatellar fat pad. Distal femur, tibial plateau, anterior/posterior femoral condyles, chamfer, and intercondylar notch cuts are performed. Trial components are placed, and alignment is checked. Synovectomy around the patellar margin is performed, with patellofemoral joint shaping and denervation. The surgical field is thoroughly irrigated. Bone cement is mixed, prostheses are implanted, and the wound is closed in layers and dressed.

   Treatment Methods:
3. Control Group: Within 24h postoperatively, anteroposterior and lateral knee X-rays are taken to confirm proper prosthesis placement. Patients are instructed to perform knee function rehabilitation exercises according to the plan. Starting from the first postoperative day, patients take placebo 3g/day after breakfast, dissolved in 200ml of warm water (40-50°C), for 4 consecutive weeks.
4. TTRJ Group: Within 24h postoperatively, anteroposterior and lateral knee X-rays are taken to confirm proper prosthesis placement. Patients are instructed to perform knee function rehabilitation exercises according to the plan. Starting from the first postoperative day, patients take freeze-dried RRTJ powder 3g/day after breakfast, dissolved in 200ml of warm water (40-50°C), for 4 consecutive weeks. The freeze-dried RRTJ juice powder used is the "Jin Ci Li" brand produced by China National Pharmaceutical Group Guizhou Great Health Industry Development Co., Ltd.

Measurement Parameters:

1. Baseline Data: Gender, age, BMI, ethnicity, occupation, education level, living and residential situation, medical history, etc.
2. Intraoperative Parameters: Operation duration, anesthesia duration, intraoperative blood loss, intraoperative average heart rate and blood pressure, etc.
3. Record adverse reactions such as wound bleeding, infection, etc.
4. Oxidative Stress Markers: Superoxide dismutase (SOD) and malondialdehyde (MDA) content measured by ELISA at preoperative 24h, postoperative 24h, 72h, and 4 weeks.
5. Inflammatory Markers (4ml blood per draw): TNF-α, IL-1, IL-6 levels measured by ELISA at preoperative 24h, postoperative 24h, and 72h.
6. Visual Analogue Scale (VAS) Pain Score: Recorded at preoperative 24h, postoperative 24h, 72h, and 4 weeks during rest and activity (walking or maximum knee flexion). Patients are explained the VAS before assessment.
7. American Knee Society (AKS) Score: Recorded at preoperative 24h, postoperative 24h, 72h, and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic criteria for primary knee osteoarthritis (KOA) as defined by the "Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2019 Edition)."
* Aged between 18 and 75 years.
* No history of trauma or surgery involving the lower limbs. Scheduled to undergo total knee arthroplasty (TKA) performed by the same surgical team at the participating hospital.
* Willing to refrain from participating in any other clinical research studies for the duration of this trial.
* Agrees to adhere to the complete study treatment regimen.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Has a preoperative knee joint infection, rheumatoid arthritis, or other concurrent inflammatory or non-inflammatory joint disease.
* Has a history of any prior knee surgery (including revision procedures).
* Has diabetes mellitus with poorly controlled glucose levels (fasting blood glucose >7.2 mmol/L or 2-hour postprandial blood glucose >11.1 mmol/L).

Has severe, unstable, or uncontrolled disease of the circulatory, respiratory, or hematopoietic systems.

* Has obesity defined as a body mass index (BMI) ≥30 kg/m².
* Has a diagnosis of severe osteoporosis.
* Is pregnant or currently breastfeeding.
* Has an active psychiatric disorder or any other condition that, in the investigator's judgment, would impair the ability to provide informed consent or comply with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Oxidative Stress Markers | Preoperative 24 hours, postoperative 24 hours, postoperative 72 hours, and postoperative 4 weeks.
  Superoxide Dismutase (SOD):
  SOD activity will be measured in serum using a commercially available human-specific ELISA kit, following the manufacturer's instructions. Results are reported in U/L.
  Malondialdehyde (MDA):
  MDA concentration will be quantified in serum using a commercial ELISA kit based on the TBARS assay, following the manufacturer's protocol. Results are reported in nmol/mL or µmol/L.
Inflammatory Markers | Preoperative 24 hours, postoperative 24 hours, and postoperative 72 hour.
  Tumor Necrosis Factor-alpha (TNF-α), Interleukin-1 (IL-1), Interleukin-6 (IL-6): The concentrations of these pro-inflammatory cytokines will be measured in serum. Quantitative detection will be performed using specific, validated human ELISA kits. These cytokines are central mediators of the systemic inflammatory response; elevated levels post-surgery are associated with pain, tissue catabolism, and delayed recovery. The assay results will provide concentrations in picograms per milliliter (pg/mL).
Visual Analogue Scale (VAS) Pain Score | Preoperative 24 hours, postoperative 24 hours, postoperative 72 hours, and postoperative 4 weeks
  Assessment Method: Pain intensity will be subjectively assessed by the patient using a 100-mm horizontal line Visual Analogue Scale. The left endpoint (0 mm) is labeled "No pain," and the right endpoint (100 mm) is labeled "Worst imaginable pain." Patients will be instructed to mark a point on the line that best represents their pain intensity at that moment.
  Scoring: The distance from the "No pain" endpoint to the patient's mark is measured in millimeters, providing a score from 0 to 100. A higher score indicates greater pain intensity.
American Knee Society (AKS) Score | Preoperative 24 hours, postoperative 24 hours, postoperative 72 hours, and postoperative 4 weeks.
  Assessment Components: The AKS Score is a physician-administered assessment comprising two separate sub-scores:
  Knee Score (0-100 points): Evaluates the knee joint itself, focusing on pain (50 points), stability (25 points), and range of motion (25 points), while deducting points for flexion contracture, extension lag, and malalignment.
  Function Score (0-100 points): Evaluates the patient's functional ability, assessing walking distance (50 points) and stair climbing (50 points). The use of walking aids leads to point deductions.
  Criteria and Definition: A higher total score indicates better knee function and less impairment. The assessment will be performed by a trained orthopedic surgeon or research nurse through patient interview and physical examination. Specific criteria for pain levels, range of motion measurement using a goniometer, ligament stability tests, and observation of gait and stair navigation will be applied strictly according to the official AKS guidelines.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol